CLINICAL TRIAL: NCT02520661
Title: Paramedic Coached ED Care Transitions to Help Older Adults Maintain Their Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-1197; 2015-1197 (Other: IRB Number); R01AG050504 (NIH); A534100 (Other: UW Madison); SMPH\EMERG MED (Other: UW Madison)
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Results first posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Emergencies; Aging
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Older adults discharged from an ED to home who receive the usual processes and services.
- Care Transitions Intervention (Active Comparator): Older adults discharged from an ED to home who receive the Care Transitions Intervention.
  Interventions: Behavioral: Care Transitions Intervention

INTERVENTIONS:
Behavioral: Care Transitions Intervention — The Care Transitions Intervention uses coaches, in this case paramedics, to support patients being discharged home by transferring skills to activate patients.
  Arms: Care Transitions Intervention

SUMMARY:
The emergency department (ED) is a common source of acute illness care for older adults. Many older adults who are discharged home from the ED return within 30 days due to numerous challenges faced during the ED-to-home transition. Unless programs to improve the ED-to-home transition are identified, the health and financial costs will only increase as the older adult population doubles by 2040. This study will apply Coleman's Care Transitions Intervention to the ED-to-home transition by adapting the program to account for the unique aspects of the ED setting. The research will evaluate the process, ED use, and cost outcomes of a community-based, paramedic-coordinated Care Transitions Intervention. Upon completion, this study will provide empiric evidence regarding this innovative approach to help the rapidly growing older adult population remain healthy and independent after an ED visit.

DETAILED DESCRIPTION:
Older adults use the emergency department (ED) as an important source of acute care, making 20 million ED visits annually. Most older adults who visit the ED do not have conditions of sufficient severity to warrant hospital admission; thus, they are treated and discharged home. Unfortunately, older adults do poorly after being discharged home from the ED, with 20% having repeat ED visits within 30 days. The ED-to-home transition has been identified as a cause for these avoidable poor outcomes, but ED-focused interventions to improve this transition have had inconclusive outcomes and have suffered from feasibility, sustainability and scalability problems.

Coleman's Care Transition Intervention (CTI) has been validated to improve the hospital-to-home transition, decreasing both hospital readmissions and costs. The CTI uses coaches, usually nurses or social workers, to support patients being discharged home by transferring skills to activate patients. Applying the CTI to the ED-to-home transition is a natural extension, but it has not been evaluated in this unique and demanding setting.

In this study, the investigators will test the hypothesis that the community-based, paramedic-coordinated ED-to-home CTI will improve community-dwelling older adults' post-ED health outcomes and reduce costs. The investigators will evaluate CTI process outcomes by testing if participants randomized to the CTI demonstrate better understanding of red flags that indicate a worsening of their condition, implement medication changes more frequently, and follow up with their primary care physicians more rapidly after ED discharge, as compared to the control group. The investigators will also evaluate the effectiveness and cost-effectiveness of the CTI by testing if participants randomized to the CTI have improved Patient Activation Measure scores 30 days after discharge, have decreased frequency of ED use, and decreased health care costs within 30 days of ED discharge. Additionally, the investigators recognize that the CTI will not eliminate all repeat ED visits. Thus, they will identify factors independently associated with repeat ED visits among CTI recipients such that future programs can ensure their needs are adequately addressed.

This research will provide critical empiric evidence regarding the significant problem of poor ED-to-home transitions. By leveraging the CTI, a widely available and efficient intervention and paramedics, a highly-skilled and respected health care provider present in all communities, the investigators will apply an innovative approach to improve older adults' health following an ED visit. Through rigorous research, they will test the effectiveness and cost-effectiveness of this approach, with a specific focus on ultimate sustainability and dissemination.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥60 years
2. English speaking
3. Monroe County, New York or Dane County, Wisconsin resident
4. University of Wisconsin or University of Rochester affiliated primary care physician
5. Community dwelling (no prisoners, nursing home, assisted living residents)
6. Discharge home from the ED

Exclusion Criteria:

1. Previous study participation
2. Discharged to hospice
3. Homelessness
4. Followed by transition care team (e.g., from recent hospitalization)
5. Followed by intensive case management program
6. Emergency Severity Index 1 patients (highest acuity, as assigned by ED triage staff)
7. Unable to obtain consent from patient or proxy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1979 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish N Shah, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Rochester Medical Center, Rochester, New York
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mi R, Hollander MM, Jones CMC, DuGoff EH, Caprio TV, Cushman JT, Kind AJH, Lohmeier M, Shah MN. A randomized controlled trial testing the effectiveness of a paramedic-delivered care transitions intervention to reduce emergency department revisits. BMC Geriatr. 2018 May 3;18(1):104. doi: 10.1186/s12877-018-0792-5. PMID 29724172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single-blind randomized controlled trial conducted at three university-affiliated hospital Emergency Departments: one in Madison, Wisconsin, and two in Rochester, New York. The study was approved by institutional review boards at the University of Wisconsin and University of Rochester with written informed consent. Enrollment and data collection occurred between January 2016 and July 2019.
Pre-assignment Details: 6,102 (11.3 percent) of 53,801 patients greater than or equal to 60 years old presenting during recruitment hours were approached for the study. Primary reasons for exclusion were inpatient admission from ED, not having a primary care provider in the health system, and living in a long-term care/assisted-living facility. After additional eligibility checks and refusals, 1,979 patients (32.4 percent) were consented and randomized into the study.
Period: Overall Study
Arm/Group | Usual Care | Care Transitions Intervention
Started | 992 | 987
Removed Following Randomization (Reasons include, admitted from ED, ED stay greater than 24 hours, other ineligibility) | 124 | 99
CTI Home Visit Scheduled (CTI = Care Transitions Intervention) | 0 | 863
Participants in Dataset | 893 | 863
Participants Completing Home Visit (Intervention arm) | 0 | 726
Participants With Primary Outcome Data (ITT) (ITT = Intent to Treat) | 886 | 860
Participants With Primary Outcome Data (PP) (PP = Per Protocol) | 886 | 725
Completed | 886 | 860
Not Completed | 106 | 127
Not completed — Lost to Follow-up | 7 | 3
Not completed — Admitted from ED | 49 | 48
Not completed — ED greater than 24 hours | 29 | 38
Not completed — other ineligibility | 14 | 22
Not completed — Withdrawal by Subject | 7 | 16

BASELINE CHARACTERISTICS:
Population: 223 enrolled participants were removed following randomization, see Participant Flow
Groups:
- Usual Care: Control Group: Older adults discharged from an ED to home who receive the usual processes and services.
- Care Transitions Intervention (ITT): Older adults discharged from an ED to home, intended to receive the Care Transitions Intervention.
- Total: Total of all reporting groups
Arm/Group | Usual Care: Control Group | Care Transitions Intervention (ITT) | Total
Number analyzed (Participants) | 893 | 863 | 1756
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.10 (8.50) | 72.69 (8.65) | 72.39 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480 | 458 | 938
  Male | 413 | 405 | 818
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 12 | 27
  Not Hispanic or Latino | 878 | 851 | 1729
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 36 | 76
  White | 818 | 800 | 1618
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 19 | 40
Region of Enrollment [Number; unit: participants]
  United States | 893 | 863 | 1756
Education [Count of Participants; unit: Participants] — Number of Participants with some college or less
  Participants | 352 | 337 | 689
Marital Status [Count of Participants; unit: Participants] — Number of Participants who are not married
  Participants | 352 | 361 | 713
Number of Charlson Comorbidities [Mean (Standard Deviation); unit: Charlson Comorbidities] — Charlson Comorbidities are nineteen conditions included in an index to predict risk of death within 1 year of hospitalization for patients with specific comorbid conditions. Extracted from participant medical records.
  Charlson Comorbidities | 2.65 (1.69) | 2.79 (1.65) | 2.72 (1.67)
Number of Participants with Deficiencies in One or more ADL [Count of Participants; unit: Participants] — Activities of Daily Living (ADL) are a list of fundamental skills required for independent living such as walking, feeding, dressing, personal hygiene, toileting, or continence.
  Participants | 299 | 332 | 631
Number of Participants with Cognitive Impairment [Count of Participants; unit: Participants] — The investigators considered participants cognitively impaired if they met any of the following conditions: (1) score > 10 on the Blessed Orientation Memory Concentration Test (BOMC); (2) self-reported a diagnosis of dementia or cognitive impairment; or (3) had medical record documentation of a memory-related condition (e.g., dementia).
  Participants | 60 | 67 | 127
Number of Participants with Inadequate Health Literacy [Count of Participants; unit: Participants] — Inadequate health literacy was measured with the Brief Health Literacy Screening Tool. Total scores range from 2-20, inadequate health literacy is considered a score between 2-12.
  Participants | 98 | 116 | 214
Number of Participants with Anxiety per GAD-2 [Count of Participants; unit: Participants] — The Generalized Anxiety Disorder-2 (GAD-2) scale has a total possible range of scores from 0-6, a score of 3 or higher indicates generalized anxiety.
  Participants | 155 | 138 | 293
Number of Participants with Moderate to Severe Depression per PHQ-9 [Count of Participants; unit: Participants] — The Patient Health Questionnaire-9 (PHQ-9) scale is a measure of depression with a total possible range of scores from 0-27. A score of greater than 10 indicates moderate or greater depression.
  Participants | 95 | 94 | 189
Perceived Health Competence Score [Mean (Standard Deviation); unit: score on a scale] — Perceived Health Competence Score (PHCS) has a total possible range of score from 8-40 where higher scores indicate a stronger perception of health competency.
  score on a scale | 29.87 (5.28) | 30.31 (5.29) | 30.09 (5.29)
Number of Participants with Fair or Poor Overall Health per SF-12 [Count of Participants; unit: Participants] — The Short Form-12 (SF-12) general health item. Participants select either Excellent, Very Good, Good, Fair, Poor, or no answer.
  Participants | 181 | 174 | 355
Number of Participants Hospitalized in 30 days prior to Emergency Department (ED) study visit [Count of Participants; unit: Participants] | 43 | 47 | 90
Number of ED visits in 30 days prior to index ED visit [Mean (Standard Deviation); unit: ED visits] | 0.12 (0.40) | 0.10 (0.34) | 0.11 (0.38)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Returning to the ED Within 30 Days of the Original ED Visit
Description: The investigators included all unplanned ED use, regardless of reason, during the 30 days after discharge as abstracted from electronic medical records (with out-of-system ED use identified during participant phone surveys). The investigators constructed dichotomous variables measuring whether or not any ED visits occurred within 14 and 30 days after discharge, with the 30-day interval being the primary prespecified outcome. Control vs Intent-to-Treat vs Per Protocol population reported.
Time Frame: 30 days after emergency department discharge
Measure: Count of Participants; unit: Participants
Groups:
- Care Transitions Intervention (ITT): Older adults discharged from an ED to home intended to receive the Care Transitions Intervention.
- Care Transitions Intervention (PP): Older adults discharged from an ED to home receive the Care Transitions Intervention per protocol.
Arm/Group | Usual Care | Care Transitions Intervention (ITT) | Care Transitions Intervention (PP)
Number analyzed (Participants) | 893 | 863 | 726
Participants
  ED revisits within 14 days | 84 | 69 | 51
  ED revisits within 30 days | 113 | 103 | 81
Statistical Analysis 1: Comparison: Usual Care vs Care Transitions Intervention (ITT); treatment relevant change in number of ED visits by 14 days; Test type: Superiority; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.62 to 1.22]
Statistical Analysis 2: Comparison: Usual Care vs Care Transitions Intervention (ITT); treatment relevant change in number of ED visits by 30 days; Test type: Superiority; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.72 to 1.30]

2. Primary Outcome: Time to Any Follow up (in Person or Phone) With PCP, Specialists, or Urgent Care
Description: Follow-up visits, abstracted from participant medical records, included office visits with primary or specialty providers, telephone calls, and online patient portal messaging (excluding automated reminder messages, electronic messages that did not receive a patient response, laboratory testing, and previously scheduled outpatient procedures). Outpatient follow-up was dichotomized by whether or not any contact with outpatient providers occurred within either 7 or 30 days of discharge. This approach allowed us to differentiate follow-up occurring soon after discharge (consistent with most ED discharge instructions) from less-timely contact with outpatient clinics. To conduct a preplanned subanalysis, we also categorized all follow-up as either "in-person" or "electronic." Dichotomous variables were created for each modality at each time point as well as a combined variable representing all forms of contact. Control vs Intent-To-Treat vs Per Protocol population reported.
Time Frame: Medical records reviewed for number of participants who followed up within 7 and 30 days, augmented by participant surveys at day 4 and 30 to learn about non-University of Wisconsin hospital visits
Measure: Count of Participants; unit: Participants
Groups:
- Care Transitions Intervention (PP): Older adults discharged from an ED to home to receive the Care Transitions Intervention per protocol.
Arm/Group | Usual Care | Care Transitions Intervention (ITT) | Care Transitions Intervention (PP)
Number analyzed (Participants) | 893 | 863 | 726
Participants
  All Follow-Up within 7 Days | 657 | 664 | 561
  All Follow-Up within 30 Days | 773 | 775 | 653
  In-Person Follow-Up within 7 days | 428 | 456 | 385
  In-Person Follow-Up within 30 days | 698 | 702 | 592
  Electronic Follow-Up within 7 Days | 510 | 524 | 445
  Electronic Follow-Up within 30 Days | 659 | 646 | 548

3. Primary Outcome: Number of Participants With Urgent Care or Unplanned Hospitalizations Within 30 Days of ED Discharge
Description: Control vs Intent-to-Treat vs Per Protocol Population reported
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Care Transitions Intervention (ITT) | Care Transitions Intervention (PP)
Number analyzed (Participants) | 893 | 863 | 726
Participants
  Urgent Care Visits | 24 | 24 | 23
  Unplanned hospitalization | 46 | 45 | 30

4. Secondary Outcome: Number of Participants With Medication Changes Implemented
Description: The investigators asked participants to self-report any medication changes (starts, stops, or modifications) they had made since discharge during the 4-day survey. They had to provide the name, classification, or purpose of each medication. Medically trained researchers compared self-reported medication changes to those listed on participants' AVS discharge instructions, excluding those with "as needed" instructions. The dichotomized variable indicates whether or not the participant reported making all recommended medication changes.
Time Frame: day 4
Population: Only participants with medication-related changes on their AVS instructions were included in this analysis
Measure: Count of Participants; unit: Participants
Groups:
- Care Transitions Intervention (ITT): Older adults discharged from an ED to home with intent to receive the Care Transitions Intervention.
Arm/Group | Usual Care | Care Transitions Intervention (ITT) | Care Transitions Intervention (PP)
Number analyzed (Participants) | 236 | 233 | 186
Participants | 78 | 73 | 65

5. Secondary Outcome: Number of Participants Who Could Recall Any Specific Red Flag
Description: The discharge instructions from the ED will be abstracted for key red flags. Participants will be asked to list the red flags for which they are monitoring their condition.
Time Frame: day 4
Population: Only patients with specific red flags listed on their discharge instructions were included in this analysis (n = 1207).
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Care Transitions Intervention (ITT) | Care Transitions Intervention (PP)
Number analyzed (Participants) | 635 | 572 | 514
Participants | 225 | 225 | 215

6. Secondary Outcome: Level of Participant Activation as Measured by the Perceived Health Competence Survey
Description: Perceived Health Competence Score (PHCS) has a total possible range of scores from 8-40 where higher scores indicate a stronger perception of health competency. This is also known as the Wallston score.
Time Frame: 30 days after emergency department discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Care Transitions Intervention (ITT) | Care Transitions Intervention (PP)
Number analyzed (Participants) | 880 | 850 | 718
score on a scale | 30.54 (4.76) | 31.12 (4.71) | 31.25 (4.77)

7. Secondary Outcome: Median Cost of Healthcare Services Within 30 Days of the Original ED Visit
Time Frame: 30 days after emergency department discharge
Population: The investigators made an informed decision not to collect cost data.
Arm/Group | Usual Care | Care Transitions Intervention
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Program Satisfaction Survey Score
Description: Participants and Caregivers were surveyed for their satisfaction with the intervention, on a scale of 0-10 where 0 is the worst experience and 10 is the best experience.
Time Frame: day 1, day 30
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Family Caregiver Activation in Transitions (FCAT)
Description: The Family Caregiver Activation in Transitions survey is a series of statements about challenges commonly faced by those caring for a loved one. It is scored on a 6 point likert scale for a total possible range between 10-60, where higher scores indicate fewer challenges to care.
Time Frame: day 1, day 30
Population: Investigators did not analyze the FCAT because of reliability issues with the instrument that led them to lack confidence in the instrument.
Arm/Group | Usual Care | Care Transitions Intervention
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Number of Participants Who Died Within 30 Days of Discharge
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Care Transitions Intervention
Number analyzed (Participants) | 893 | 863
Participants | 5 | 2

ADVERSE EVENTS:
Time Frame: up to 30 days
Description: Adverse Events data reported for all participants who were randomized for study. MedDRA System Order Class (SOC) reported for all adverse events and serious adverse events.
Arm/Group | Usual Care | Care Transitions Intervention
All-Cause Mortality (participants affected / at risk) | 5/992 | 2/987
Serious Adverse Events (participants affected / at risk) | 51/992 | 51/987
Other Adverse Events (participants affected / at risk) | 93/992 | 76/987
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=992) | Care Transitions Intervention (N=987)
Blood and Lymphatic Disorders (Blood and lymphatic system disorders) | 1 | 0
Cardiac Disorders (Cardiac disorders) | 7 | 11
Gastrointestinal Disorders (Gastrointestinal disorders) | 8 | 6
General Disorders (General disorders) | 3 | 2
Infections and Infestations (Infections and infestations) | 4 | 6
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 | 0
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 7 | 3
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous System Disorders (Nervous system disorders) | 4 | 6
Renal and urinary disorders (Renal and urinary disorders) | 3 | 4
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Vascular disorders (Vascular disorders) | 3 | 4
Surgical and Medical Procedures (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=992) | Care Transitions Intervention (N=987)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 1
Cardiac Disorders (Cardiac disorders) | 13 | 7
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 | 1
Endocrine Disorders (Endocrine disorders) | 0 | 2
Gastrointestinal Disorders (Gastrointestinal disorders) | 9 | 10
General Disorders (General disorders) | 7 | 5 — There is one 'unknown' event counted in this category.
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 0
Immune System Disorders (Immune system disorders) | 1 | 0
Infections and Infestations (Infections and infestations) | 4 | 3
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 7 | 8
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 3 | 4
Musculoskeletal and connective tissues disorders (Musculoskeletal and connective tissue disorders) | 10 | 6
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nervous System Disorders (Nervous system disorders) | 9 | 5
Psychiatric disorders (Psychiatric disorders) | 3 | 1
Renal and Urinary Disorders (Renal and urinary disorders) | 4 | 2
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 | 0
Surgical and Medical procedures (Surgical and medical procedures) | 3 | 1
Vascular Disorders (Vascular disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT02520661/Prot_SAP_000.pdf